CLINICAL TRIAL: NCT01361737
Title: Serum Markers in Preeclamptic Women
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Oslo University Hospital, Rikshospitalet, OsloUH
Other Study IDs: NOSERPE11
Record Dates: First submitted 2011-05-25; First posted 2011-05-27 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2011-05

CONDITIONS: Preeclampsia
Keywords: Preeclampsia; serological bio-bank; adiponectin; suPAR
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- preeclampsia: * Control group: 86 healthy women not developing preeclampsia (PE)
  * Case group: 43 women developing PE

SUMMARY:
Could possible markers in serum obtained in the first trimester predict the human-pregnancy specific disorder pre-eclampsia?

ELIGIBILITY:
Inclusion Criteria:

* previous healthy

Exclusion Criteria:

* Previous inflammatory diseases

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Norwegian pregnant women
Sampling Method: Probability Sample
Dates: Start 1999-01; Primary Completion 1999-01 (Actual); Study Completion 2004-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Rikshospitalet, Oslo, Norway